CLINICAL TRIAL: NCT05373576
Title: Neurofunctional Correlates of the Behavioral Modifications Associated With Tachidino in Children With Developmental Dyslexia
Acronym: TACHIDINO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 877
Record Dates: First submitted 2022-05-04; First posted 2022-05-13 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Dyslexia, Developmental
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACHIDINO (Experimental)
  Interventions: Behavioral: TACHIDINO
- WAITING LIST (No Intervention)

INTERVENTIONS:
Behavioral: TACHIDINO — TACHIDINO is based on two principles a) selective stimulation of a cerebral hemisphere and specific reading strategies, and b) the training of selective visuospatial attention, as well as the perception of rapid movement and the visual characteristics of words even in the presence of so-called visual crowding or "crowding", an automatic effect of our perceptual system that leads to "obfuscation" of the visual areas surrounding the object to be analyzed, to make its vision clearer (as suggested by the "Magnocellular theory" of dyslexia; Stein et al., 2019).
  Arms: TACHIDINO

SUMMARY:
Developmental dyslexia (DD) is the most common learning disorder. Multiple cognitive and sensory domains contribute to the etiology of DD and develop before reading acquisition. Atypical brain functional responses and structural features have been found in the reading developing circuitry. Treatments addressing visual-spatial attention and motion perception (Visual Attention Training; VAT) are among the most effective interventions in Italian children with DD. The VAT seems to improve the efficiency of the visual attention system and the magnocellular (M) pathway which is crucial for learning to read. Evidence for impaired M function in subjects with DD in the visual striate and extra-striate cortex have been reported. How these treatments affect the brain functionality is still not clear. Since DD has a neurobiological basis, it is important to deeply investigate atypical functional responses and structural features in reading-related areas, and to understand how treatments operate at the neuronal level. A growing number of studies investigates structural and functional measures in neurodevelopmental disorders by using high-resolution MRI at high field (3T and 7T). Similarly, several studies examine the effects of different types of reading training upon brain activity. Better understanding of the relationship between structural/functional abnormalities and DD could disentangle the causes of reading difficulties and helps in developing effective treatments.

The significance of this study is twofold: 1) NEURAL CORRELATES OF TREATMENT: The investigators expect TACHIDINO to specifically affect the underlying neurophysiological functioning which influences reading skills in children with DD; 2) BRAIN SIGNATURES: As integrated multi-domain data (behavioral and brain imaging) are complementary to each other, they could enhance the possibility to find unique treatment/brain functioning combinations to evaluate the effectiveness of intervention and to predict the treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Reading skills (both accuracy and speed) below -2.00 standard deviation

Exclusion Criteria:

* No ADHD
* No contraindications to magnetic resonance

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain activation as assessed by fMRI | baseline
  BOLD signal in regions of interest (ROIs) underlying reading network
Brain activation as assessed by fMRI | before the intervention
  BOLD signal in regions of interest (ROIs) underlying reading network
Brain activation as assessed by fMRI | immediately after the intervention
  BOLD signal in regions of interest (ROIs) underlying reading network

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS Eugenio Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No